CLINICAL TRIAL: NCT06032442
Title: An Open Randomized Prospective Study of the Supporting Properties of the Dietary Supplement ARTNEO in Comparison With Active Control in Parallel Groups in Patients With Knee Osteoarthritis Aged 40 to 75 Years
Brief Title: A Study to Assess Efficacy of Supporting Properties and Safety of ARTNEO in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ArtNeo-terra
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis; Osteo Arthritis Knee; Osteoarthritis, Knee
Keywords: undenatured type ii collagen; collagen; Boswellia serrata; methylsulfonylmethane; osteoarthritis; knee pain
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — hydroquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARTNEO (Experimental): 1 capsule 1 time per day for 6 months
  Interventions: Dietary Supplement: ARTNEO
- Artra (Active Comparator): 1 tablet 2 times per day for 6 months
  Interventions: Drug: Artra

INTERVENTIONS:
Dietary Supplement: ARTNEO — Dietary Supplement: undenatured collagen type II, methylsulfonylmethane, boswellia serrata, vitamin D3 (cholecalciferol), vitamin C (ARTNEO)
  Release form: capsules with an average weight of 585 mg. Active ingredients: MCM (methylsulfonylmethane) 300 mg, vitamin C (ascorbic acid) 80 mg, boswellia extract (65% boswellic acids) 50.05 mg, undenatured (native) type II collagen 40 mg, vitamin D3 (cholecalciferol) 400 IU.
  Suggested Use: Adults, 1 capsule daily with meals.
  Arms: ARTNEO
Drug: Artra — Active ingredients:
  Glucosamine hydrochloride 500 mg Chondroitin sulfate sodium 500 mg
  Excipients:
  dibasic calcium phosphate, microcrystalline cellulose, croscarmellose sodium, stearic acid, magnesium stearate.
  Orally; adults and children over 15 years of age are prescribed 1 tablet 2 times a day for the first three weeks; 1 tablet 1 time per day for the next weeks and months.
  Arms: Artra

SUMMARY:
The goal of the interventional study is to assess the effectiveness of the supporting properties and safety of the dietary supplement ARTNEO (ARTNEO®), capsules with an average weight of 585 mg, in patients with osteoarthritis of the knee joint of both sexes aged 40 to 75 years. The main questions it aims to answer are:

1. To evaluate the effectiveness of the supporting properties of dietary supplement ARTNEO (ARTNEO®) in patients with knee osteoarthritis in comparison with active control;
2. To evaluate the safety of the dietary supplement ARTNEO (ARTNEO®) in patients with knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent to participate in the study
* Men and women aged 40-75 years old, able to move independently, BMI 18-35 kg/m2
* Verified osteoarthritis involving the target knee according to the American College of Rheumatology (ACR) criteria at least 3 months prior to study entry, i.e. pain in the knee joint in combination with one of the following signs: crepitus in the joint or morning stiffness in the joint lasting less than 30 minutes in association with radiographic findings in the target knee joint
* X-ray stage I-III osteoarthritis in the target knee joint according to the Kellgren-Lawrence classification with a predominant lesion of the medial tibiofemoral area of the knee joint (X-ray of the target knee joint during the screening period or within 6 months prior to the screening visit)
* Regular associated pain in the target knee joint within the last 3 months
* Pain severity from 45 to 74 mm (moderate pain) on 100 mm VAS in the target knee joint after a washout screening period and confirmation of a 48-hour complete abstinence from rescue therapy (pain in motion (when starting a movement and walking around the office))
* Lequesne score of 5-7 for the joint being assessed after a washout screening period and confirmation of 48 hours of complete abstinence from rescue therapy;
* The ability to understand the rules of the study, the willingness to follow them, as well as the ability and ability to go through the procedures provided for in the study;
* Willingness to avoid the use of ibuprofen, aspirin (>100 mg/day), and other NSAIDs or other pain medications (OTC and prescription) other than paracetamol as a "rescue drug" throughout the study (maximum dosage allowed per protocol) 1,500 mg per day, with a complete withdrawal required 48 hours before Visits 2 - 6 and Visit 9)
* Willingness to refuse complementary and alternative medicine therapy, as well as willingness to restrict diet (excluded soy, avocado, passion fruit, pineapple, turmeric, foods enriched with ω-3 fatty acids, decoction of willow bark, pine, mugwort, L-carnitine, acupuncture and etc.)
* Women of childbearing potential must have a negative pregnancy test at screening (except women who have had a hysterectomy or who have gone through menopause for more than 2 years)

Exclusion Criteria:

* Pregnancy, lactation or planning pregnancy during the study period
* Individual intolerance to the active or excipients of the dietary supplement ARTNEO (non-denatured type II collagen + methylsulfonylmethane + Boswellia serrata extract + vitamin C + Vitamin D3), the reference drug and the "rescue drug" paracetamol (acetaminophen)
* Intolerance to eggs, poultry, shellfish;
* History of trauma or surgery on the target knee joint (other than diagnostic arthroscopy more than 60 days old at study entry), expected surgery (within 6 months following inclusion)
* Positive test results for HIV, viral hepatitis B or C, syphilis.
* Diseases that, from the point of view of the investigator, put the patient's health at risk if participating in the study or potentially make it difficult to interpret the results of the study (may affect the assessment of endpoints)
* Known or suspected malignancy at the time of screening or in the previous 2 years, other than completely healed skin cancer in situ;
* Immune-inflammatory joint disease, systemic connective tissue disease, or severe osteoarthritis (target joint after washout screening period and 48-hour complete withdrawal of rescue drug, motion VAS score > 74 mm and/or Lequesne score > 7 points), systemic red lupus
* History of gout
* Diseases of the gastrointestinal tract: enteritis, colitis, Crohn's disease, irritable bowel syndrome, ulcerative colitis and any other diseases of the gastrointestinal tract, which, in the doctor's opinion, may affect the absorption and assimilation of the active components of the drugs, in particular, the formation of the mechanism of oral immunotolerance to undenatured collagen
* Hemophilia and other hemorrhagic diathesis, as well as taking anticoagulants and antiplatelet agents
* Fibromyalgia and other chronic pain syndromes
* Impaired kidney function (GFR less than 60 ml / min / 1.73 m2 as assessed by the Cockcroft-Gault formula at the screening visit), severe chronic renal failure
* Severe liver dysfunction (ALT, AST levels 3 times or more above the upper limit of normal, and / or total bilirubin level 1.5 times or more above the upper limit of normal)
* Mental and / or neurological diseases with partial or complete loss of legal capacity
* Presence or suspicion of drug, alcohol or drug addiction
* Intra-articular injection in the target knee joint:

  1. Hyaluronates - less than 6 months prior to randomization
  2. Other high molecular weight synovial fluid prostheses in less than 24 months
  3. Glucocorticosteroids - less than 1 month prior to randomization visit
  4. NSAIDs less than 3 weeks before randomization
* The need for stable use of glucocorticosteroids in any dosage form
* Failure to comply with the washout screening period and 48 hours of complete withdrawal of the rescue drug (immediately prior to baseline measurement at Visit 2, Day 1) in relation to prohibited therapy, in particular the use of paracetamol, ibuprofen, aspirin or other NSAIDs, any pain medication in any drug form, as well as some natural products (such as soy, avocado, passion fruit, pineapple, turmeric, products enriched with ω-3 fatty acids, decoction of willow bark, pine, wormwood), L-carnitine
* Use of glucocorticosteroids, SYSADOA (Symptomatic Slow-Acting Drugs in Osteoarthritis) in the period of 3 months before randomization
* Use of ω-3 polyunsaturated fatty acid preparations in the 6 months prior to randomization (a 2-week washout period is allowed), therapeutic doses of fish or vegetable oils (≥ 2 g/day), shark cartilage preparations
* Participation in another clinical study at present or in the previous 30 days or 5 half-lives (whichever is longer) prior to the Screening Visit
* History of treatment with oral undenatured type II collagen or anti-tumor necrosis factor (TNF) antibodies

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Change in the mean of the total score on The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale | Baseline to month 6
  Change in total WOMAC score at Visit 9 (day 180 ± 4) from baseline at Visit 2 (day 1)

SECONDARY OUTCOMES:
Change in mean WOMAC total score (baseline to day 7, months 1 and 3) | Baseline to day 7, months 1 and 3
  Change in mean WOMAC total score at Visit 3 (Day 7 ± 2), Visit 4 (Day 30 ± 2), Visit 6 (Day 90 ± 3) from baseline at Visit 2 (Day 1)
Change in the mean on the subscales of the WOMAC (scales of pain, stiffness, functional insufficiency) | Baseline to day 7, months 1, 3, 6
  Change in the mean score on subscales of the WOMAC scale (pain, stiffness, functional impairment scale) at Visit 3 (Day 7 ± 2), Visit 4 (Day 30 ± 2), Visit 6 (Day 90 ± 3) and Visit 9 (Day 180) ± 4) compared to baseline at Visit 2 (Day 1)
Change in the mean score on the Lequesne scale | Baseline to day 7, months 1, 3, 6
  Change in the mean score on the Lequesne scale (gonarthrosis severity index) at Visit 3 (day 7 ± 2), at Visit 4 (day 30 ± 2), Visit 6 (day 90 ± 3) and Visit 9 (day 180 ± 4) by compared to baseline (at Visit 2, Day 1)
Evaluation of magnetic resonance imaging (MRI) signs of damage to the target joint | Baseline to month 6
  Evaluation of MRI signs of damage to the target joint according to the MRI protocol, including the parameters "synovial thickness", "thickness of the intra-articular effusion", "bone marrow edema", "cartilage changes" at Visit 9 (day 180 ± 4) compared with baseline at Visit 2 (Day 1).
Change in mean 100-mm visual analogue scale (VAS) in the target knee joint | Baseline to day 7, months 1, 2, 3, 6
  Change in mean 100-mm VAS score at the target knee (pain in motion: at the start of the movement and while walking around the office) at Visit 3 (Day 7 ± 2), Visit 4 (Day 30 ± 2), Visit 5 (Day 60) ± 2), Visit 6 (day 90 ± 3) and Visit 9 (day 180 ± 4) compared to baseline at Visit 2 (day 1).
  VAS scores range from 0 ("no pain") to 100 ("the worst pain imaginable").
Changing the circumference of the target knee joint | Baseline to months 1, 3, 6
  Change in target knee circumference at Visit 4 (Day 30 ± 2), Visit 6 (Day 90 ± 3), and Visit 9 (Day 180 ± 4) from baseline at Visit 2 (Day 1)
Change in the paracetamol intake | Baseline to day 7, months 1, 2, 3, 6
  Patient diary assessment of total number of paracetamol tablets (500 mg dosage) taken since Day 1 (Visit 2, Day 1) and change in the number of patients (%) reporting consumption at Visit 3 (Day 7 ± 2), Visit 4 (Day 30 ± 2), Visit 5 (Day 60 ± 2), Visit 6 (Day 90 ± 3) and Visit 9 (Day 180 ± 4) compared to baseline at Visit 2 (Day 1);
The number of cases of dropping out of patients (%) due to the ineffectiveness of therapy | Baseline to month 6
  The number of patients dropping out (%) due to the need to prescribe non-steroidal anti-inflammatory drugs (NSAIDs) and other pain medications (with the exception of paracetamol rescue drug at prescribed doses) or due to the need to increase the dose allowed under the protocol (1,500 mg per day: 3 tablets per day). 500 mg) paracetamol
Change in the mean score on the The Short Form-36 (SF-36) quality of life questionnaire | Baseline to months 1, 3, 6
  Change in Mean SF-36 Quality of Life Score at Visit 4 (Day 30 ± 2), Visit 6 (Day 90 ± 3), and Visit 9 (Day 180 ± 4) from Baseline at Visit 2 (Day 1).
  SF-36 results in eight domain scores. Each of them ranges from 0 to 100% with 100% indicating the best result possible.
Evaluation of the effectiveness of therapy by a doctor on the Integrative Medicine Outcome Scale (IMOS) | Baseline to month 6
  Evaluation of the effectiveness of therapy by a doctor at the end of the course of treatment (IMOS scale).
  Score ranges from 0 to 4 with 0 indicating the best result: complete recovery (0 points), significant improvement (1 point), slight to moderate improvement (2 points), no change (3 points), worsening (4 points).
Evaluation of the effectiveness of ongoing therapy by the patient according to the Integrative Medicine Outcome Scale (IMOS) scale | Baseline to month 6
  Evaluation of the effectiveness of the therapy by the patient on the IMOS scale.
  Score ranges from 0 to 3 with 0 indicating the best result: excellent (0 points), good (1 point), satisfactory (2 points), not effective (3 points).

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Mazurov, MD, Principal Investigator — North-Western State Medical University named after I.I.Mechnikov
Locations (1):
- Federal State Budgetary Educational Institution of Higher Education "North-Western State Medical University named after I.I. Mechnikov" of the Ministry of Health of Russia, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: No